CLINICAL TRIAL: NCT01269853
Title: Phase I/II Trial Of Repeated Super-selective Intraarterial Cerebral Infusion Of Bevacizumab (Avastin) for Treatment of Relapsed/Refractory Glioblastoma Multiforme and Anaplastic Astrocytoma.
Brief Title: Repeated Super-selective Intraarterial Cerebral Infusion of Bevacizumab (Avastin) for Treatment of Relapsed GBM and AA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Professor, Feinstein Institute for Medical Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-353
Record Dates: First submitted 2010-12-22; First posted 2011-01-04 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: GBM; AA; AO; Brain; Tumors; Malignant; Glioblastoma; Multiforme; Anaplastic; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Experimental)
  Interventions: Drug: Bevacizumab
- Arm 1 (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Experimental portion of this proposal:
  This trial will have two experimental arms that will be open labeled and non-randomized.
  ARM 1 (If the patient has multifocal disease or leptomeningeal disease)
  Day 0: Intraarterial Bevacizumab single dose (15mg/kg) after Mannitol to open the blood brain barrier Day 28: Intravenous Bevacizumab (10mg/kg) every two weeks thereafter until disease progression on MRI scan.
  If progression occurs, repeat Intraarterial Bevacizumab single dose (15mg/kg) to area of progression and wait 28 days and then restart Intravenous Bevacizumab (10mg/kg) every two weeks thereafter until progression on MRI scan.
  Repeat Cycle
  Arms: Arm 2
Drug: Bevacizumab — ARM 2 (If the patient has no multifocal disease or leptomeningeal disease)
  Day 0: Intraarterial Bevacizumab single dose (15mg/kg) after Mannitol to open the blood brain barrier Day 28: No biweekly IV Bevacizumab treatment
  If MRI shows progression then repeat Intraarterial Bevacizumab single dose (15mg/kg) to area of progression Repeat Cycle
  Arms: Arm 1

SUMMARY:
The high-grade malignant brain tumors, glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA), comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival durations of only 9-12 months for GBM, and 3-4 years for AA. Initial therapy consists of either surgical resection, external beam radiation or both. All patients experience a recurrence after first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. It is unknown if currently used intravenous (IV) therapies even cross the blood brain barrier (BBB). The investigators have shown in a previous phase I trial that a single Super-selective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab (up to 15mg/kg) is safe and effective in the treatment of recurrent GBM. Therefore, this phase I/II clinical research trial is an extension of that trial in that the investigators seek to test the hypothesis that repeated dosing of intraarterial Bevacizumab is safe and effective in the treatment of recurrent malignant glioma. By achieving the aims of this study the investigators will also determine if IV therapy with Bevacizumab should be combined with repeated selected intraarterial Bevacizumab to improve progression free and overall survival. The investigators expect that this project will provide important information regarding the utility of repeated SIACI Bevacizumab therapy for malignant glioma, and may alter the way these drugs are delivered to the patients in the near future.

DETAILED DESCRIPTION:
The current standard of care for recurring GBM is for patients to receive Bevacizumab (Avastin) intravenously (IV) at 10mg/kg every two weeks until their tumor grows more than 25%. At that point, these patients are deemed treatment failures and are given another treatment. Because of the blood brain barrier (BBB) where IV drugs do not penetrate the blood vessel walls well to get into the brain, no one knows for sure if these IV drugs actually get into the brain after infusion. We have recently completed a Phase I clinical trial that has shown that SIACI of Bevacizumab is safe and effective up to a dose of 15mg/kg in patients with recurrent malignant glioma. This two arm open-label, non-randomized trial is a follow up study to that trial and will ask two simple questions: Is it safe to deliver repeated doses of Bevacizumab intraarterially using these super selective intraarterial delivery techniques? Is it necessary to combine this IA regimen of treatment with biweekly IV Bevacizumab in order to improve progression free survival (PFS) and overall survival (OS)? Information from this trial will yield important answers to the durability and efficacy of this delivery technique and may radically change the way chemotherapy is given to our patients with brain tumors.

Current Standard of Care:

Day 0: Intravenous Bevacizumab (10mg/kg) Day 14, 28 (and every two weeks thereafter): Intravenous Bevacizumab

Therefore the experimental aspects of this treatment plan will include:

1. Subjects will first be treated with Mannitol prior to chemotherapy infusion (Mannitol 20%; 12.5 mL/s over 2 minutes) in order to disrupt the blood brain barrier. This technique has been used in several thousand patients in previous studies for the IA delivery of chemotherapy for malignant glioma. We have used this without complication in the 30 patients from our Phase I protocol as well.
2. To treat patients with one of two arms with repeated intraarterial delivery (SIACI) of Bevacizumab for patients with recurring or relapsing high grade glioma. Each arm gets IA delivery with one arm getting IV Bevacizumab biweekly as well and the other arm not getting intervening IV therapy. In each arm, IA therapy is repeated when MRI shows progression. Persistent progression after three intraarterial chemotherapies would remove the patient from the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Patients with a documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA) or anaplastic mixed oligoastrocytoma (AOA).
* Patients must have at least one confirmed and evaluable tumor site. A confirmed tumor site is one in which is biopsy-proven.
* Patients must have a Karnofsky performance status 70% (or the equivalent ECOG level of 0-2).
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period.

Exclusion Criteria:

* Previous treatment with greater than 2 cycles of Bevacizumab at 10mg/kg (2 IV Infusions).
* Women who are pregnant or lactating.
* Patients with significant inter-current medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2010-10; Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Composite overall response rate (CORR) | 6 months
  We will determine this composite overall response rate (CORR) through the Response Assessment in Neuro-Oncology (RANO) criteria
Progression-free survival (PFS) and overall survival (OS) | 6 month
  Six-month progression-free survival (PFS) and overall survival (OS) will be assessed by Kaplan-Meier survival analysis, assuming adequate follow-up time

SECONDARY OUTCOMES:
The safety of repeated SIACI of mannitol and Bevacizumab at 15mg/kg. | 1 month
  The descriptive frequency of subjects experiencing toxicities will also be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States